CLINICAL TRIAL: NCT04231747
Title: A Phase 1, Multicenter, Open-label Study of CC-97540, CD19-targeted NEX-T Chimeric Antigen Receptor (CAR) T Cells, in Subjects With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A Study of CC-97540, CD19-targeted NEX-T Chimeric Antigen Receptor (CAR) T Cells, in Subjects With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-97540-NHL-001; U1111-1244-9049 (Registry Identifier: UTN)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma Non-Hodgkin; Agressive Lymphoma; Diffuse-large B-cell Lymphoma (DLBCL)
Keywords: Lymphoma; B-cell non-Hodgkin lymphoma; Agressive Lymphoma; Diffuse-large B-cell Lymphoma; DLBCL; NHL; CC-97540; CD19; NEX-T chimeric antigen receptor (CAR) T cells; CAR-T; CART
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Dendritic Cell Sarcoma, Interdigitating; Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-97540 monotherapy (Experimental): Subjects will be assigned to receive CC-97540 followed by 3 consecutive doses of lymphodepleting chemotherapy (fludarabine IV (30 mg/m2/day) and cyclophosphamide IV (300 mg/m2/day).
  Interventions: Biological: CC-97540

INTERVENTIONS:
Biological: CC-97540 — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to produce CC 97540.
  During CC 97540 production, subjects may receive bridging chemotherapy for disease control. Upon successful generation of CC 97540 product, subjects will receive treatment with CC 97540 therapy.
  Each cycle will include lymphodepleting chemotherapy followed by one dose of CC 97540 administered by intravenous (IV) injection.

SUMMARY:
This is a Phase 1, first-in-human, open-label, multicenter study of CC-97540, CD19-targeted NEX-T chimeric antigen receptor (CAR) T cells, in subjects with relapsed or refractory B-cell non-Hodgkin lymphoma.

The study will consist of 2 parts: dose-escalation (Part A) and dose-expansion (Part B). The dose-escalation part (Part A) of the study is to evaluate the safety and tolerability of increasing dose levels of CC-97540 to establish a recommended Phase 2 dose (RP2D); and the dose-expansion part (Part B) of the study is to further evaluate the safety, pharmacokinetics/pharmacodynamics, and efficacy of CC-97540 at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Age ≥ 18 years at the time of informed consent.
2. Signed written informed consent obtained prior to any study procedure.
3. Willing and able to adhere to the study visit schedule and other protocol requirements.
4. Relapsed and/or refractory aggressive B-cell NHL as defined:

   1. Histologically confirmed DLBCL not otherwise specified, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (HGBCL), transformed DLBCL from follicular (tFL) or marginal zone lymphoma (tMZL), primary mediastinal B-cell lymphoma (PMBCL), or FL grade 3b (FL3B) (Note: Subjects with Richter's transformation (transformed DLBCL from CLL) are ineligible) AND
   2. Have relapsed and/or refractory disease after at least 2 lines of systemic therapy which must include at least one anthracycline and rituximab (or other anti-CD20 monoclonal antibody).

      Note: Lines of therapy will exclude those given for prior indolent lymphoma. It is not required for subjects to have had anthracycline for their DLBCL if received for indolent disease AND/OR
   3. Have relapsed and/or refractory DLBCL failed to ASCT treatment. Note: ASCT failure is defined as either failure to achieve an objective response (PR or better), or disease progression after ASCT(Note: Subjects who were not candidates to receive ASCT treatment (due to age or other factors) are eligible; the reason for not receiving ASCT must be documented in the electronic case report form (eCRF).
5. Positron emission tomography (PET)-positive disease as per the Lugano Classification (at screening or following bridging therapy, whichever is later).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate organ function as detailed in the protocol.
8. Adequate vascular access for leukapheresis.
9. Willing and able to undergo tumor biopsies (in subjects with accessible disease).
10. Agree to not donate blood, organs, sperm or semen, and egg cells for usage in other individuals as detailed in the protocol.
11. Female and male subjects agree to use effective contraception as detailed in the protocol.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the Investigator; or unwillingness or inability to follow the procedures required in the protocol.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Central nervous system (CNS)-only involvement by malignancy (note: subjects with pathologically-confirmed secondary CNS involvement are allowed).)
5. Prior CAR T- cell or genetically-modified T- cell therapy, or prior CD19- targeted therapy (including, but not limited to, anti-CD19 mAbs or bispecific antibodies).)
6. Treatment with the following therapies or procedure within the specified period:

   1. Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) within 14 days before leukapheresis administration. Physiologic replacement, topical, and inhaled steroids are permitted.
   2. Cytotoxic chemotherapeutic agents (eg, doxorubicin, vincristine, gemcitabine, oxaliplatin, carboplatin, etoposide) within 7 days of leukapheresis, with the exception of alkylating agents.
   3. Intrathecal therapy (eg, dexamethasone, methotrexate, cytosine arabinoside, cytarabine) within 7 days of leukapheresis.
   4. Oral chemotherapeutic agents, including lenalidomide and ibrutinib, are allowed if at least 5 half-lives have elapsed prior to leukapheresis.
   5. Alkylating agents (eg, cyclophosphamide, ifosfamide, bendamustine) within 4 weeks of leukapheresis.
   6. Any experimental therapy within 8 weeks (for biologics) or 5 half-lives (for small molecules) before leukapheresis
   7. Immunosuppressive therapies within 4 weeks of leukapheresis (eg, calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate, rapamycin, immunosuppressive antibodies such as anti-TNF, anti-IL6, or anti-IL6R)
   8. Monoclonal antibodies (including rituximab, polatuzumab, etc.) within 7 days.
   9. Donor lymphocyte infusions within 6 weeks of leukapheresis
   10. Radiation within 6 weeks of leukapheresis. Subjects must have progressive disease in irradiated lesions or have additional non-irradiated, PET-positive lesions to be eligible. Radiation to a single lesion, if additional non-irradiated PET-positive lesions are present, is allowed up to 14 days prior to leukapheresis.
   11. Autologous stem-cell transplant (SCT) (ie, Day 0 receipt of hematopoietic stem cells) within 3 months of leukapheresis
   12. Washout of prior therapy (eg, bridging therapy for disease control)
7. Active autoimmune disease requiring immunosuppressive therapy.
8. Allogenic SCT (ie, Day 0 receipt of hematopoietic stem cells) within 6 months of leukapheresis or presence of ongoing symptoms or treatment for chronic graft-versus host disease (GVHD).)
9. Hypersensitivity to fludarabine and/or cyclophosphamide.
10. Prior history of malignancies, other than studied NHL, unless the subject has been free of the disease for ≥ 2 years except for the following non-invasive malignancies:

    1. Basal or squamous cell carcinoma of the skin
    2. Carcinoma in situ of the cervix or the breast
    3. Incidental histologic finding of prostate cancer (T1a or T1b using the TNM (tumor, nodes, metastasis) clinical staging system) or prostate cancer that is curative
    4. Other completely resected stage 1 solid tumor with low risk for recurrence
11. Active hepatitis B, hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening.
12. Uncontrolled or active systemic fungal, bacterial, viral or other infection despite appropriate anti-infection treatment at the time of leukapheresis or pre-treatment evaluation.
13. History of any one of the following cardiovascular conditions within the 6 months prior to screening: Class III or IV heart failure as defined by the New York Heart Association, myocardial infarction, unstable angina, angioplasty or stenting, or other clinically significant cardiac disease.
14. History or presence of clinically significant CNS pathology such as seizure disorder, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, or cerebellar disease. Presence of clinically active psychosis.
15. History of ≥ Grade 2 hemorrhage within 30 days of screening.
16. Pregnant or nursing (lactating) women.
17. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to leukapheresis or initiation of LD chemotherapy.

    -Acute symptoms must have resolved and based on investigator assessment in consultation with the Sponsor Medical Monitor, there are no sequelae that would place the subject at a higher risk of receiving study treatment.
18. Previous SARS-CoV-2 vaccine within 14 days prior to leukapheresis or initiation of LD chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From the time of informed consent and follow up to 2 years after infusion of CC-97540
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.ject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the sub

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to 2 years after CC-97540 infusion
  The proportion of subjects with a best overall response of complete response (CR).
Overall response Rate (ORR) | Up to 2 years after CC-97540 infusion
  The proportion of subjects achieving CR or partial response (PR).
Duration of response (DOR) | Up to 2 years after CC-97540 infusion
  The time from first response to progressive disease (PD) or death.
Time to response (TTR) | Up to 2 years after CC-97540 infusion
  Time from CC-97540 infusion to the first documentation of response (CR or PR).
Time to complete response (TTCR) | Up to 2 years after CC-97540 infusion
  Time from CC-97540 infusion to the first documentation of CR
Progression free survival (PFS) | Up to 2 years after CC-97540 infusion
  Time from CC-97540 infusion to the first documentation of PD, or death from any cause, whichever occurs first
Overall survival (OS) | Up to 2 years after CC-97540 infusion
  Time from CC-97540 infusion to death
Pharmacokinetics - peak expansion (Cmax) | Up to 2 years after CC-97540 infusion
  Maximum blood concentration
Pharmacokinetics -time to peak expansion (tmax) | Up to 2 years after CC-97540 infusion
  Time to peak (maximum) blood concentration
Pharmacokinetics - elimination half-life (t1/2) | Up to 2 years after CC-97540 infusion
  Elimination half-life
Pharmacokinetics - Area under curve (AUC) | Up to 2 years after CC-97540 infusion
  Area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (11):
  - Local Institution - 003, Birmingham, Alabama
  - Local Institution - 004, Atlanta, Georgia
  - Local Institution - 011, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Nebraska Medicine Fred and Pamela Buffett Cancer Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Local Institution - 001, New York, New York
  - Local Institution - 008, New York, New York
  - Local Institution - 010, Charlotte, North Carolina
  - Oregon Health and Science University OHSU, Portland, Oregon
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah
- Canada (3):
  - Foothills Medical Centre - Tom Baker Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04231747.html